CLINICAL TRIAL: NCT03937986
Title: Influence of Orexin Antagonism on Motivation for Cocaine
Brief Title: Suvorexant and Cocaine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BED IN 39; R01DA048617 (NIH)
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — suvorexant; Cocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Subjects will be maintained on oral placebo. Cocaine will be administered acutely during placebo maintenance. Placebo will be administered acutely during placebo maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo oral capsule
- Suvorexant Dose 1 (Experimental): Subjects will be maintained on oral suvorexant dose 1. Cocaine will be administered acutely during suvorexant dose 1 maintenance. Placebo will be administered acutely during suvorexant dose 1 maintenance.
  Interventions: Drug: Suvorexant; Drug: Cocaine
- Suvorexant Dose 2 (Experimental): Subjects will be maintained on oral suvorexant dose 2. Cocaine will be administered acutely during suvorexant dose 2 maintenance. Placebo will be administered acutely during suvorexant dose 2 maintenance.
  Interventions: Drug: Suvorexant; Drug: Cocaine
- Suvorexant Dose 3 (Experimental): Subjects will be maintained on oral suvorexant dose 3. Cocaine will be administered acutely during suvorexant dose 3 maintenance. Placebo will be administered acutely during suvorexant dose 3 maintenance.
  Interventions: Drug: Suvorexant; Drug: Cocaine

INTERVENTIONS:
Drug: Suvorexant — The pharmacodynamic effects of suvorexant maintenance will be determined.
  Arms: Suvorexant Dose 1; Suvorexant Dose 2; Suvorexant Dose 3
Drug: Cocaine — The pharmacodynamic effects of cocaine will be determined during maintenance on placebo and suvorexant.
Drug: Placebo oral capsule — The pharmacodynamic effects of placebo will be determined.
  Arms: Placebo

SUMMARY:
The research proposed here will translate findings from preclinical research and provide the initial clinical evidence that orexin antagonism reduces motivation for cocaine, as well as other cocaine-associated maladaptive behaviors in active cocaine users. This study will also provide basic science information about the orexinergic mechanisms underlying the pharmacodynamic effects of cocaine in humans. As such the outcomes will contribute to our understanding of the clinical neurobiology of cocaine use disorder. Overall, the proposed work seeks to expand the scope of current clinical neuroscience research on cocaine addiction by focusing on orexin, which has strong preclinical evidence supporting its critical role in addiction but remains unstudied in humans.

ELIGIBILITY:
Inclusion Criteria:

* Recent cocaine use

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance abuse or dependence that are deemed by the study physicians to interfere with study completion
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation
* Females not currently using effective birth control
* Contraindications to cocaine, methylphenidate or duloxetine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W Stoops, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Included in Analysis: This study used a within subjects design (i.e., all subjects were to receive all oral suvorexant maintenance conditions [0, 5, 10 and 20 mg] and intravenous cocaine doses [0, 10 and 30 mg/70 kg]). Seven subjects completed the full study. An eighth was enrolled but discharged at the outset of the COVID-19 pandemic. Data from completed sessions for that subject are included here.
Period: Overall Study
Arm/Group | Subjects Included in Analysis
Started | 8
Completed | 7
Not Completed | 1
Not completed — COVID-19 Pandemic | 1

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Included in Analysis
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Reinforcing Effects of Cocaine
Description: Number of Times Subjects Choose Cocaine (Maximum of 10 Choices) Over Money
Time Frame: 12 times over approximately 1 month inpatient admission.
Measure: Mean (Standard Error); unit: Number of Cocaine Choices
Groups:
- Dose Condition 1: 0 mg/70 kg IV Cocaine and 0 mg/day Oral Suvorexant
- Dose Condition 2: 10 mg/70 kg IV Cocaine and 0 mg/day Oral Suvorexant
- Dose Condition 3: 30 mg/70 kg IV Cocaine and 0 mg/day Oral Suvorexant
- Dose Condition 4: 0 mg/70 kg IV Cocaine and 5 mg/day Oral Suvorexant
- Dose Condition 5: 10 mg/70 kg IV Cocaine and 5 mg/day Oral Suvorexant
- Dose Condition 6: 30 mg/70 kg IV Cocaine and 5 mg/day Oral Suvorexant
- Dose Condition 7: 0 mg/70 kg IV Cocaine and 10 mg/day Oral Suvorexant
- Dose Condition 8: 10 mg/70 kg IV Cocaine and 10 mg/day Oral Suvorexant
- Dose Condition 9: 30 mg/70 kg IV Cocaine and 10 mg/day Oral Suvorexant
- Dose Condition 10: 0 mg/70 kg IV Cocaine and 20 mg/day Oral Suvorexant
- Dose Condition 11: 10 mg/70 kg IV Cocaine and 20 mg/day Oral Suvorexant
- Dose Condition 12: 30 mg/70 kg IV Cocaine and 20 mg/day Oral Suvorexant
Arm/Group | Dose Condition 1 | Dose Condition 2 | Dose Condition 3 | Dose Condition 4 | Dose Condition 5 | Dose Condition 6 | Dose Condition 7 | Dose Condition 8 | Dose Condition 9 | Dose Condition 10 | Dose Condition 11 | Dose Condition 12
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 7 | 7 | 8 | 8 | 7 | 7 | 7 | 7
Number of Cocaine Choices | 1.3 (3.5) | 5.0 (5.3) | 8.3 (3.) | 0 (0) | 3.7 (8.4) | 8.4 (2.7) | 1.3 (3.5) | 8.1 (3.7) | 9.3 (1.9) | 0.4 (1.1) | 6.6 (4.7) | 8.7 (1.9)

ADVERSE EVENTS:
Time Frame: 32 months
Description: Definitions for adverse events/serious adverse events follow clinicaltrials.gov guidelines.
Arm/Group | Subjects Included in Analysis
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Included in Analysis (N=8)
Elevated Heart Rate (Cardiac disorders) | 1
Elevated Blood Pressure (Cardiac disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 1
Burning Sensation (Skin and subcutaneous tissue disorders) | 1
IV Needle Infiltration (Skin and subcutaneous tissue disorders) | 1
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1
Hand Swelling (Skin and subcutaneous tissue disorders) | 2
Arm Soreness (Skin and subcutaneous tissue disorders) | 1
Saline Taste from IV Flush (Gastrointestinal disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Increased Dream Activity (Nervous system disorders) | 1
Increased Sleep (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT03937986/Prot_SAP_000.pdf